CLINICAL TRIAL: NCT03698032
Title: Pistachios as a Recovery Food Following Rigorous Exercise in Trained Athletes
Brief Title: Effect of Pistachios on Muscle Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Mark Kern, Professor, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: S00022068
Record Dates: First submitted 2018-10-01; First posted 2018-10-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Muscle Soreness
MeSH Terms: conditions — Myalgia | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water Arm (Active Comparator): Participants will consume water only as the intervention
  Interventions: Dietary Supplement: Water
- 1.5 oz Pistachios (Active Comparator): Participants will consume water plus 1.5 oz of pistachios as the intervention
  Interventions: Dietary Supplement: 1.5 oz Pistachios
- 3.0 oz Pistachios (Active Comparator): Participants will consume water plus 3.0 oz of pistachios as the intervention
  Interventions: Dietary Supplement: 3.0 oz Pistachios

INTERVENTIONS:
Dietary Supplement: Water — Participants will consume water only
  Arms: Water Arm
Dietary Supplement: 1.5 oz Pistachios — Participants will consume water plus 1.5 oz of pistachios as the intervention
  Arms: 1.5 oz Pistachios
Dietary Supplement: 3.0 oz Pistachios — Participants will consume water plus 3.0 oz of pistachios as the intervention
  Arms: 3.0 oz Pistachios

SUMMARY:
Pistachios are an understudied and often unappreciated functional food. While nuts in general have received somewhat more attention for their nutritional properties from researchers, practitioners and the media, pistachios often seem to be overlooked. Meanwhile, pistachios appear to possess characteristics that suggest that they are likely to impart benefits that are equal to and perhaps above and beyond those of average nuts. We intend to explore the potential impacts of pistachios on recovery from rigorous exercise in well-trained athletes. We hypothesize that feeding 1.5 oz of pistachios will improve exercise recovery as determined by a reduction in delayed onset muscle soreness and suppression of markers of muscle damage, inflammation and oxidative stress in comparison to water and that the benefits will be greater with consumption of 3.0 oz of pistachios.

DETAILED DESCRIPTION:
Specific objectives are to determine the dose response to ingestion of pistachios for promotion of recovery from vigorous exercise. To accomplish this, investigators will examined whether regular consumption of pistachios followed by pistachio feeding at two different doses (1.5 and 3.0 oz) during the recovery period following eccentrically biased exercise (downhill running) promotes enhanced recovery as measured by muscle soreness, markers of muscle damage, and status for inflammation and oxidative stress in comparison to a control feeding of water in endurance-trained runners (18-35 years of age).

Study Design

A cross-over design performed in random order will be utilized in which participants will complete 3 trials separated by at least 3-4 weeks. At each testing site, 28 well-trained, competitive male athletes will be recruited. Participants will be required to participate in at least 5 hours of vigorous exercise per week and to actively compete in sport. Exclusion criteria include smoking, medications known to impact inflammation, musculoskeletal limitations and use of supplements known to impact antioxidant or inflammatory status within 1 month of participation.

Approach/Methods

Participants will consume water only, water plus 1.5 oz of pistachios, or water plus 3.0 oz of pistachios daily for 2 weeks during 3 separate trials in a randomized, cross-over fashion. Subjects will then report to the laboratory following an overnight fast and after abstaining from strenuous exercise for 2 days. Fasting blood samples will be collected and participants will complete a 40-min downhill run at -10% grade at 65-70% of a predetermined VO2max. A recovery serving of water or water along with one of the doses of pistachios will be provided. Antecubital blood samples will be collected before the bout of exercise and 24, 48, and 72 hours afterward. Muscle soreness will be assessed at each timepoint as well. Vertical jump will be assessed prior to the exercise bout and at each recovery timepoint. Daily consumption of the pistachios will continue during the 72-hour recovery period.

All participants will receive individualized diet counseling by investigators on a biweekly basis. An initial 3-day food record will be analyzed using dietary software to serve as a starting point for which the diet counseling will be based. Each participant will be provided with an individualized plan outlining their required macronutrient and micronutrient intakes (including antioxidants) in grams corresponding to their habitual diet as determined by the 3-day diet diary. Once per week, participants will provide a 3-day food record to track compliance with the nutrition protocol. All participants will be provided with feedback in their next biweekly private counseling session. To ensure that the results were due, as much as possible, to the differing dietary intervention (pistachio ingestion), participants will be instructed not to take any vitamin or mineral supplements during the study.

Data will be analyzed using a repeated measures ANOVA followed by paired T-tests as post-hoc tests using SPSS. Statistical significance will accepted at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* 28 well-trained
* Competitive male athletes
* Must participate in at least 5 hours of vigorous exercise per week
* Must actively compete in sport.

Exclusion Criteria:

* Smoking
* Medications known to impact inflammation
* Medications known to impact musculoskeletal limitations
* Use of supplements known to impact antioxidant or inflammatory status within 1 month of participation

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
change from baseline of serum creatine kinase at 24, 48 and 72 hours | before the bout of exercise and 24, 48, and 72 hours afterward
  Serum will be analyzed for concentrations of creatine kinase as marker of muscle damage

SECONDARY OUTCOMES:
Change from baseline of serum c-reactive protein at two weeks | Baseline and after two weeks of test food consumption
  For change in inflammatory response
Change from baseline of body weight at two weeks | Baseline and after two weeks of test food consumption

CONTACTS AND LOCATIONS:
Locations (1):
- San Diego State University, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rayo VU, Thayer I, Galloway SDR, Hong MY, Hooshmand S, Liu C, North E, Okamoto L, O'Neal T, Philpott J, Witard OC, Kern M. Influence of pistachios on force production, subjective ratings of pain, and oxidative stress following exercise-induced muscle damage in moderately trained athletes: A randomized, crossover trial. Metabol Open. 2022 Oct 21;16:100215. doi: 10.1016/j.metop.2022.100215. eCollection 2022 Dec. PMID 36325128